CLINICAL TRIAL: NCT04766515
Title: Multicenter Observational Prospective Study of Immune Checkpoint Inhibitors in Patients With Solid Neoplasms
Brief Title: Observational Prospective Study of Immune Checkpoint Inhibitors for Solid Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Other Study IDs: ARION
Record Dates: First submitted 2021-02-20; First posted 2021-02-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective, multicenter observational study included all patients with solid neoplasms who received treatment with immune checkpoint inhibitors (ICIs) in clinical practice, regardless of tumor type, tumor stage, type of immunotherapy, or treatment lines. This study aimed to assess the use, effectiveness, and safety of ICIs for solid neoplasms in real-world populations, which can provide insights into clinical decisions associated with the use of ICIs for the treatment of cancer patients in the real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years.
* Pathologically confirmed diagnosis of a solid tumor cancer.
* Patients receiving treatment with immune checkpoint inhibitors.
* Ability to understand and willingness to provide the informed consent.

Exclusion Criteria:

* Age < 18 years.
* Patients with hematological malignancies or solid benign tumors.
* Mental disorders, drug abuse, and social condition that may negatively impact compliance in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with solid tumors treated with immune-checkpoints inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Three years
  OS was defined as the time from the date of first administration of immunotherapy until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.

SECONDARY OUTCOMES:
Progression Free Survival | Three years
  PFS was measured from the date of first administration of immunotherapy to the date of disease progression as defined by Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 or death due to any cause, whichever occurred first. For patients whose disease did not progress, PFS was evaluated by censoring patients at their most recent imaging.
Overall Objective Response Rate | At least 6 weeks after start of treatment
  ORR was defined as the proportion of participants with partial response (PR) or complete response (CR) to treatment as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Percentage of Participants With Adverse Events | Three years
  Treatment-related adverse events were assessed and graded according to CTCAE v. 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengfei Zhu, MD, Principal Investigator — Fudan University; Qian Chu, MD, Study Director — Tongji Hospital; Jie Hu, MD, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Dong H, Lan A, Gao J, An Y, Chu L, Yang X, Chu X, Hu J, Chu Q, Ni J, Zhu Z. Prognostic significance of bone metastasis and clinical value of bone radiotherapy in metastatic non-small cell lung cancer receiving PD-1/PD-L1 inhibitors: results from a multicenter, prospective, observational study. Transl Lung Cancer Res. 2024 Oct 31;13(10):2603-2616. doi: 10.21037/tlcr-24-441. Epub 2024 Oct 18. PMID 39507037